CLINICAL TRIAL: NCT03806946
Title: Impact of Relationship of Epilepsy and Attention Deficit Hyperactive Disorder
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, Assistent lecture, Assiut University
Other Study IDs: Impact of ADHD and epilepsy
Record Dates: First submitted 2018-05-09; First posted 2019-01-16 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Attention-Deficit Hyperactivity Disorder; Epilepsy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Epilepsy | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- group1: ADHD with normal EEG
  Interventions: Diagnostic Test: electroencephalography; Diagnostic Test: psychometric scales to diagnosis psychiatric disorders; Other: psychometric scales for assesment socioeconomic and behaviour problems
- group 2: ADHD with abnormal EEG
  Interventions: Diagnostic Test: electroencephalography; Diagnostic Test: psychometric scales to diagnosis psychiatric disorders; Other: psychometric scales for assesment socioeconomic and behaviour problems
- group 3: Epilepsy
  Interventions: Diagnostic Test: electroencephalography; Diagnostic Test: psychometric scales to diagnosis psychiatric disorders; Other: psychometric scales for assesment socioeconomic and behaviour problems
- group 4: Healthy control group
  Interventions: Diagnostic Test: electroencephalography; Diagnostic Test: psychometric scales to diagnosis psychiatric disorders; Other: psychometric scales for assesment socioeconomic and behaviour problems
- group 5: ADHD and epilepsy
  Interventions: Diagnostic Test: electroencephalography; Diagnostic Test: psychometric scales to diagnosis psychiatric disorders; Other: psychometric scales for assesment socioeconomic and behaviour problems

INTERVENTIONS:
Diagnostic Test: electroencephalography — diagnosis epileptic discharge
  Other Names: EEG
Diagnostic Test: psychometric scales to diagnosis psychiatric disorders — to diagnosis intellectual disability, attention deficit hyperactivity disorder ,epilepsy,autism and other mental illness.
  Other Names: WISC III (Wechsler Intelligence Scale for Children),conners 3rd Edition,(cbcl)The Child Behavior Checklis,Epilepsy interview,The Childhood Autism Spectrum Test (CAST)
Other: psychometric scales for assesment socioeconomic and behaviour problems — to assessment other behavioural comorbidity as aggression ,mood changes,etc and help in identify function impairment, social and economic burden
  Other Names: socioeconomic class, pediatric quality of life inventory, The Strengths and Difficulties Questionnaire (SDQ),The Mood and Feelings Questionnaire (MFQ),

SUMMARY:
The most common neuropsychiatric disorder in early childhood is attention deficit/hyperactivity disorder (ADHD) with evidence of abnormality in structure and function of brain. Epilepsy is one of the commonest comorbidity associated with ADHD with negative outcome on childrens' quality of life, and is considered to be a risk for academic underachievement. These two disorders are highly associated, with more possibility to be a bidirectional relationship. The mechanisms of this comorbidity are unknown. In this association, a difficult challenge is presented since antiepileptic therapy and drugs used to treat ADHD may aggravate the clinical picture of each other. The main objectives are to evaluate this overlap of those disorders, find their complications on child and his family, and to suggest possible solutions to improve the outcome of those children.

DETAILED DESCRIPTION:
The commonest childhood disorder is attention deficit hyperactivity disorder(ADHD) which continues into adulthood.The main two symptoms are inattention and hyperactivity.

As epilepsy is one of the commonest comorbidity with ADHD to about (40%), there are many overlap symptoms between both disorders for example:

* Behavioral features which are shared in both frontal lobe epilepsy with ADHD such as impulsivity, disinhibition, and irritability
* The electroencephalogram: there is an increase in the rate of spikes in children with ADHD with no epileptic symptoms, which supports the theory of presence similar mechanism about central nervous system dysfunction.

These reasons lead to increase obstacles for diagnosis, assessment, and treatment for both disorders.

As this comorbidity duplicates the complications (i.e. drop the school, financial cost, stress on families, negative effect on academic, vocational, social relations and self-esteem ) so there is a great need to study this comorbidity to give a proper care for these patients.

In this study, all participants will be enrolled over a period of 12 months from Assiut outpatients clinic .All participants will be assessed in the psychiatric interview by using prepared child and adolescent psychiatric sheet include (psychiatric and neurology history, physical examination and mental state examination). After that electroencephalogram(EEG) will be done to diagnoses epilepsy and identify different types of seizures.

All participants will be categorizing into 4 groups ( ADHD, epilepsy, ADHD,and epilepsy, healthy) according to EEG and the psychiatric sheet. Each group will be assessed by different psychometrics scales to evaluate cognitive, social, economic and behavioral outcome. The results of all groups will be analysed by using Stata version 15 to evaluate the effect of ADHD and epilepsy in children and adolescent and identify the possible risk factors to improve outcome

ELIGIBILITY:
Inclusion Criteria:

* Both males and females were included.
* Age range from 6- 11 years.
* Diagnosis of ADHD and/or epilepsy was verified and confirmed either on a clinical basis or by using reliable psychometric tests.
* In epilepsy groups: only Idiopathic type was included.
* Willing of the parents or the caregivers to participate in the study.

Exclusion Criteria:

* Children whom caretakers refused to give informed consent.
* Children with intelligence quotient below 70.
* Children with history or current substance use.
* Children with medical or other neurological conditions.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: childern and adolescent attending psychiatric outpatients clinic of Assiut university who had diagnosis of attention deficit hyperactivity disorder or epilepsy or both and with age (6y-11y)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
measure intellectual equations for children with epilepsy and ADHD | baseline
  WISC-III provided scores for Verbal IQ (VIQ), Performance IQ (PIQ), and Full-Scale IQ (FSIQ).
  The child's verbal IQ score was derived from scores on six of the subtests: information, digit span, vocabulary, arithmetic, comprehension, and similarities.
  The child's performance IQ was derived from scores on the remaining seven subtests: picture completion, picture arrangement, block design, object assembly, coding, mazes, and symbol search.
  The overall intelligence quotient, called the full scale IQ, as well as a verbal IQ and a performance IQ. The three IQ scores are standardized in such a way that a score of 100 is considered average and serves as a benchmark for higher and lower scores.
measure socioeconomic class for families and children with comorbid epilepsy and ADHD | baseline
  It will be measure by Socioeconomic class scale which consist of It contain four main variables 1-the educational level of the father and mother 2-the occupation of the father and mother 3-total family income 4-life style of the family. The total score of the scale equal the sum of scores in each level, the scores 36-42 mean the high socioeconomic class, the scores 21-26 mean the low socioeconomic class, and scores between them mean the middle class.
measure mood and feeling changes in children with comorbid epilepsy and ADHD. | baseline
  It will be measure by Mood and Feelings Questionnaire (MFQ) arent Report is a 13-item measure assessing recent depressive and describe feelings and mood,more than 26 is consider for evaluation of depression
measure quality of life for children with comorbid epilepsy and ADHD | baseline
  It is composed of 23 items that assessment function in the following four areas: physical (eight items), emotional (five items), social (five items), and school (five items). Patients report their function using a 5-point Likert scale ranging from 0 to 4. These responses are reverse scored and linearly transformed to a 0 to 100 scale, with a higher score indicating a higher QOL.
  The Psychosocial Health Summary score is a computed mean of the emotional, social, and school functioning subscales of the PedsQL. The physical functioning scale is the same as the Physical Summary score. In addition, the computed mean of the Emotional, Social, School functioning, and Physical scales are used to generate a Total Summary score. PedsQL scales are composed of parallel child self-report and parent-proxy report formats.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-Din Darweesh, PhD, Study Director — Assiut University; HossamEddin Ahmad, PhD, Study Chair — Assiut University; Patrick Bolton, PhD, Study Chair — King's College London
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Result] Dunn DW, Austin JK, Huster GA. Behaviour problems in children with new-onset epilepsy. Seizure. 1997 Aug;6(4):283-7. PMID 9304719
- [Result] Kanner AM. The use of psychotropic drugs in epilepsy: what every neurologist should know. Semin Neurol. 2008 Jul;28(3):379-88. doi: 10.1055/s-2008-1079342. Epub 2008 Jul 24. PMID 18777484
- [Result] Chou IC, Chang YT, Chin ZN, Muo CH, Sung FC, Kuo HT, Tsai CH, Kao CH. Correlation between epilepsy and attention deficit hyperactivity disorder: a population-based cohort study. PLoS One. 2013;8(3):e57926. doi: 10.1371/journal.pone.0057926. Epub 2013 Mar 6. PMID 23483944
- [Result] Sherman EM, Slick DJ, Connolly MB, Eyrl KL. ADHD, neurological correlates and health-related quality of life in severe pediatric epilepsy. Epilepsia. 2007 Jun;48(6):1083-91. doi: 10.1111/j.1528-1167.2007.01028.x. Epub 2007 Mar 22. PMID 17381442
- [Result] Kaufmann R, Goldberg-Stern H, Shuper A. Attention-deficit disorders and epilepsy in childhood: incidence, causative relations and treatment possibilities. J Child Neurol. 2009 Jun;24(6):727-33. doi: 10.1177/0883073808330165. PMID 19491115
- [Result] Kirov R, Kinkelbur J, Banaschewski T, Rothenberger A. Sleep patterns in children with attention-deficit/hyperactivity disorder, tic disorder, and comorbidity. J Child Psychol Psychiatry. 2007 Jun;48(6):561-70. doi: 10.1111/j.1469-7610.2007.01729.x. PMID 17537072
- [Result] Dickstein, L.J., Roba, M.B. and Oldham, J.M.(1997): Review of psychiatry. AmericanPsychiatric Press. Washington, DC. London,England.
- [Derived] Ahmed GK, Darwish AM, Khalifa H, Khashbah MA. Evaluation of psychiatric comorbidity in attention-deficit hyperactivity disorder with epilepsy: A case-control study. Epilepsy Res. 2021 Jan;169:106505. doi: 10.1016/j.eplepsyres.2020.106505. Epub 2020 Nov 21. PMID 33302225